CLINICAL TRIAL: NCT02345226
Title: A Phase 3b, Randomized, Double-Blind Study to Evaluate Switching From a Regimen Consisting of Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF) Fixed Dose Combination (FDC) to Emtricitabine/Rilpivirine/ Tenofovir Alafenamide (FTC/RPV/TAF) FDC in Virologically-Suppressed, HIV-1 Infected Subjects
Brief Title: Study to Evaluate Switching From a Regimen Consisting of Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate (EFV/FTC/TDF) Fixed Dose Combination (FDC) to Emtricitabine/Rilpivirine/Tenofovir Alafenamide (FTC/RPV/TAF) FDC in Virologically-Suppressed, HIV-1 Infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-366-1160; 2014-004779-21 (EudraCT Number)
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: HIV-1 Infection
Keywords: HIV
MeSH Terms: interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FTC/RPV/TAF (Experimental): FTC/RPV/TAF plus EFV/FTC/TDF placebo for at least 96 weeks.
  Interventions: Drug: FTC/RPV/TAF; Drug: EFV/FTC/TDF Placebo
- EFV/FTC/TDF (Active Comparator): EFV/FTC/TDF plus FTC/RPV/TAF placebo for at least 96 weeks.
  Interventions: Drug: EFV/FTC/TDF; Drug: FTC/RPV/TAF Placebo
- Open Label Extension Phase (Experimental): After the Week 96 visit, participants will be given the option to receive open label FTC/RPV/TAF for up to an additional 48 weeks. In countries where FTC/RPV/TAF is not yet commercially available, participants will be given the option to receive open-label FTC/RPV/TAF and attend visits every 12 weeks until FTC/RPV/TAF becomes commercially available, or until Gilead elects to discontinue the study, whichever occurs first.
  Interventions: Drug: FTC/RPV/TAF

INTERVENTIONS:
Drug: FTC/RPV/TAF — 200/25/25 mg FDC tablets administered orally once daily
  Other Names: Odefsey®
  Arms: FTC/RPV/TAF; Open Label Extension Phase
Drug: EFV/FTC/TDF Placebo — Tablets administered orally once daily
  Arms: FTC/RPV/TAF
Drug: EFV/FTC/TDF — 600/200/300 mg FDC tablets administered orally once daily
  Other Names: Atripla®
  Arms: EFV/FTC/TDF
Drug: FTC/RPV/TAF Placebo — Tablets administered orally once daily
  Arms: EFV/FTC/TDF

SUMMARY:
The primary objective of this study is to evaluate the non-inferiority of switching to emtricitabine/rilpivirine/tenofovir alafenamide (FTC/RPV/TAF) fixed dose combination (FDC) as compared to continuing the non-nucleoside reverse transcriptase inhibitor (NNRTI) regimen of efavirenz /FTC/tenofovir disoproxil fumarate (EFV/FTC/TDF) FDC in virologically-suppressed HIV-1 infected participants.

ELIGIBILITY:
Key Inclusion Criteria:

* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Currently receiving EFV/FTC/TDF FDC for ≥ 6 consecutive months preceding the screening visit
* Documented plasma HIV-1 RNA levels < 50 copies/mL (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is > 50 copies/mL) for ≥ 6 months preceding the screening visit. Unconfirmed virologic elevation of ≥ 50 copies/mL after previously reaching viral suppression (transient detectable viremia, or "blip") and prior to screening is acceptable
* Have no documented resistance to any of the study agents at any time in the past
* HIV-1 RNA < 50 copies/mL at the screening visit
* Hepatic transaminases (AST and ALT) ≤ 5 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm^3; platelets ≥ 50,000/mm^3; hemoglobin ≥ 8.5 g/dL)
* Serum amylase ≤ 5 × ULN (individuals with serum amylase > 5 × ULN will remain eligible if serum lipase is ≤ 5 × ULN)
* Normal ECG (or if abnormal, determined by the Investigator to be not clinically significant)
* Adequate renal function: Estimated glomerular filtration rate ≥ 50 mL/min according to the Cockcroft-Gault formula

Key Exclusion Criteria:

* Hepatitis B surface antigen (HBsAg) positive
* Hepatitis C antibody positive with detectable hepatitis C virus (HCV) RNA (individuals who have HCV antibody but no detectable HCV RNA are eligible to enroll)
* Individuals experiencing or with a medical history of decompensated cirrhosis (e.g., ascites, encephalopathy, etc.)
* Females who are breastfeeding
* Positive serum pregnancy test
* Current alcohol or substance use judged by the Investigator to potentially interfere with the individual's study compliance
* A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma. Individuals with cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of Baseline/Day 1 and must not be anticipated to require systemic therapy during the study
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Baseline/Day 1
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements
* Participation in any other clinical trial (including observational trials) without prior approval from the sponsor is prohibited while participating in this trial
* Individuals receiving ongoing therapy with any of the disallowed medications listed in the protocol, including drugs not to be used with FTC, RPV and/or TAF; or individuals with any known allergies to the excipients of FTC/RPV/TAF

Note: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2015-01-26 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2019-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (117):
- United States (79):
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Spectrum Medical Group, Phoenix, Arizona
  - AHF Research Center, Beverly Hills, California
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Long Beach Education and Research Consultants, Long Beach, California
  - Kaiser Permanente, Los Angeles, California
  - Southern California Men's Medical Group, Los Angeles, California
  - Tarrant County ID Associates, Los Angeles, California
  - Kaiser Permanente, Sacramento, California
  - University of California-UC Davis, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - Optimus Medical, San Francisco, California
  - Kaiser Permanente, San Leandro, California
  - Los Angeles BioMedical Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Apex Research Institute, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - World Health Clinicians' CIRCLE CARE Center, Norwalk, Connecticut
  - Capital Medical Associates, P.C., Washington D.C., District of Columbia
  - Medical Faculty Associates, Inc., Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - AIDS Healthcare Foundation, Miami, Florida
  - University of Miami, Miami, Florida
  - AIDS Healthcare Foundation, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Diseases Associates of NW Florida, P.A., Pensacola, Florida
  - Hillsborough County Health Dept., Tampa, Florida
  - Infectious Disease Research Institute Inc., Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - AIDS Research & Treatment Center of the Treasure Coast, Vero Beach, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Rowan Tree Medical PA, Wilton Manors, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Atlanta ID Group, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - The CORE Foundation, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Boston University Medical Center, Boston, Massachusetts
  - Brigham and Women's, Boston, Massachusetts
  - MetroWest Medical Center, Framingham, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Upstate Infectious Diseases Associates, Albany, New York
  - North Shore University Hospital, Manhasset, New York
  - Columbia University Medical Center/ New York Presbyterian, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Infectious Disease Consultants, PA, Charlotte, North Carolina
  - The Brody School of Medicine, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - Trinity Health and Wellness Center/AIDS Arms, Inc., Dallas, Texas
  - AIDS Arms, Inc./Trinity Health & Wellness Center, Fort Worth, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
  - Peter Shalit, MD, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
- Belgium (2):
  - CHU Saint-Pierre University Hospital, Brussels
  - Cliniques Universitaires UCL Saint-Luc, Brussels
- Canada (8):
  - University of Alberta, Edmonton, Alberta
  - Spectrum Health, Vancouver, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Maple Leaf Research, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Clinique medicale l'Actuel, Montreal, Quebec
  - Clinique OPUS, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- France (3):
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Saint Louis, Paris
  - Chu Tours, Tours
- Germany (9):
  - Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH (zibp), Berlin
  - University of Bonn, Bonn
  - Universitat zu Koln, Cologne
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Infektiologikum, Frankfurt
  - ICH Study Center Hamburg, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - MUC Research GmbH, München
- Puerto Rico (3):
  - Clinical Research Puerto Rico Inc, San Juan
  - Hope Clinical Research, San Juan
  - University of Puerto Rico School of Medicine, San Juan
- Spain (6):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic i Provincial, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitary de Bellvitge, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Switzerland (3):
  - University Hospital Basel, Basel
  - Geneva University Hospital, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- United Kingdom (4):
  - Barts & The London NHS Trust, London
  - King's College Hospital, London
  - Mortimer Market Centre, London
  - The Royal Free Hampstead NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and transparency
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Hagins D, Orkin C, Daar ES, Mills A, Brinson C, DeJesus E, Post FA, Morales-Ramirez J, Thompson M, Osiyemi O, Rashbaum B, Stellbrink HJ, Martorell C, Liu H, Liu YP, Porter D, Collins SE, SenGupta D, Das M. Switching to coformulated rilpivirine (RPV), emtricitabine (FTC) and tenofovir alafenamide from either RPV, FTC and tenofovir disoproxil fumarate (TDF) or efavirenz, FTC and TDF: 96-week results from two randomized clinical trials. HIV Med. 2018 Nov;19(10):724-733. doi: 10.1111/hiv.12664. Epub 2018 Aug 12. PMID 30101539
- [Result] Mills A, Brinson C, Martorell C, Crofoot G, Daar E, Osiyemi O, et al. Switching to RPV/FTC/TAF from RPV/FTC/TDF or EFV/FTC/TDF: Week 96 Results. Conference on Retroviruses and Opportunistic Infections, Boston. March 4-7, 2018, Abstract 504.
- [Result] Arribas JR, Rockstroh J, Post, Yazdanpanah Y, Cavassini, DeJesus E, et al. Bone and renal safety of switching to rilpivirine/emtricitabine/tenofovir alafenamide (RPV/FTC/TAF) from single-tablet regimens (STRs) containing efavirenz/emtricitabine/tenofovir disoproxil fumarate (EFV/FTC/TDF) or rilpivirine/emtricitabine/tenofovir disoproxil fumarate (RPV/FTC/TDF): Week 48 subgroup analysis in patients at risk of or with comorbidities. Abstract accepted for presentation at the 16th European AIDS Conference, 2017 25-27 October Milan, Italy.
- [Result] Porter DP, KulkarniR, Cao H, SenGupta D, and White KL. No Emergent Resistance in HIV-1 Virologically-Suppressed Subjects Who Switched to RPV/FTC/TAF [Poster 1381]. ID Week 2017 4-8 October; San Diego, California.
- [Result] E DeJesus, M Ramgopal, G Crofoot, P Ruane, A LaMarca. J-M Molina et al. Efficacy and Safety of Switching to RPV/FTC/TAF in Older Adults. 8th International Workshop on HIV and Aging 2017 2-3 October, New York, New York.
- [Result] Molina JM, DeJesus E, Rijnders B, Post FAV, B., Stoeckle M, ThalmeA, et al. Efficacy and Safety of Switching From RPV/FTC/TDF or EFV/FTC/TDF to RPV/FTC/TAF in Black Adults [Presentation MOPEB0291]. 9th IAS Conference on HIV Science 2017 23-26 July Paris, France.
- [Result] Rockstroh J, Orkin C, Yazdanpanah Y, Di Perri GDS, P. E., Arribas JR, Brinkman K, et al. Switching From TDF to TAF Improves Bone and Renal Safety Independent of Age, Sex, Race, or 3rd Agent: Results From Pooled Analysis (N=3816) of Virologically Suppressed HIV-1 Infected Adults [Presentation MOPEB0289]. 9th IAS Conference on HIV Science; 2017 23 26 July Paris, France.
- [Result] DeJesus E, Ramgopal M, Crofoot G, Ruane P, LaMarca A, Mills A, Martorell CT, de Wet J, Stellbrink HJ, Molina JM, Post FA, Valero IP, Porter D, Liu Y, Cheng A, Quirk E, SenGupta D, Cao H. Switching from efavirenz, emtricitabine, and tenofovir disoproxil fumarate to tenofovir alafenamide coformulated with rilpivirine and emtricitabine in virally suppressed adults with HIV-1 infection: a randomised, double-blind, multicentre, phase 3b, non-inferiority study. Lancet HIV. 2017 May;4(5):e205-e213. doi: 10.1016/S2352-3018(17)30032-2. Epub 2017 Mar 2. PMID 28259776
- [Result] Majeed SR, Shao Y, Garner W, Scott J, Pérez-Ruixo C, SenGupta D, et al. Evaluation of RPV/FTC/TAF Exposure-Efficacy and Exposure-Safety Relationships [Poster 427]. Conference on Retroviruses and Opportunistic Infections (CROI) 2017 13-16 February; Seattle, Washington.
- [Result] Hagins D, Mills A, Martorell C, Walmsley S, Gallant J, Tebas P, et al. Efficacy and Safety of Switching to RPV/FTC/TAF in Women [Abstract 12]. 7th International Workshop on HIV & Women; 2017 11-12 February; Seattle, Washington.
- [Result] Orkin C, DeJesus E, Ramgopal M, Crofoot G, Ruane P, LaMarca A, et al. 48 Week Results from two studies: Switching to RPV/FTC/TAF from EFV/FTC/TDF (Study 1160) or RPV/FTC/TDF (Study 1216) [Presentation]. HIV Glasgow; 2016 23-26 October; Glasgow, United Kingdom.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe and North America. The first participant was screened on 26 January 2015. The last study visit occurred on 02 January 2019.
Pre-assignment Details: 974 participants were screened.
Groups:
- FTC/RPV/TAF: Double-Blind Phase: Emtricitabine/rilpivirine/tenofovir alafenamide (FTC/RPV/TAF) (200/25/25 mg) fixed-dose combination (FDC) tablet + efavirenz/emtricitabine/tenofovir disoproxil fumarate (EFV/FTC/TDF) placebo tablet orally once daily for up to 96 weeks.
  Open-Label Extension Phase: After the Week 96 visit, participants were given the option to receive open label FTC/RPV/TAF FDC for up to an additional 48 weeks. In countries where FTC/RPV/TAF FDC was not yet commercially available, participants were given the option to receive open-label FTC/RPV/TAF FDC orally once daily and attend visits every 12 weeks until FTC/RPV/TAF FDC became commercially available, or until Gilead elected to discontinue the study, whichever occurred first.
- EFV/FTC/TDF: Double-Blind Phase: EFV/FTC/TDF (600/200/300 mg) FDC tablet + FTC/RPV/TAF placebo tablet orally once daily for up to 96 weeks.
  Open-Label Extension Phase: After the Week 96 visit, participants were given the option to receive open label FTC/RPV/TAF FDC for up to an additional 48 weeks. In countries where FTC/RPV/TAF FDC was not yet commercially available, participants were given the option to receive open-label FTC/RPV/TAF FDC orally once daily and attend visits every 12 weeks until FTC/RPV/TAF FDC became commercially available, or until Gilead elected to discontinue the study, whichever occurred first.
Period: Double-Blind Phase
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Started | 440 | 441
Completed | 371 | 370
Not Completed | 69 | 71
Not completed — Adverse Event | 5 | 6
Not completed — Death | 3 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Investigator's Discretion | 4 | 3
Not completed — Non-Compliance with Study Drug | 1 | 2
Not completed — Withdrew Consent | 41 | 39
Not completed — Lost to Follow-up | 12 | 16
Not completed — Randomized but Never Treated | 2 | 4
Period: Open-Label Extension Phase
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Started | 25 (346 participants completed the Double-Blind Phase, but did not enter Open-Label Extension Phase.) | 21 (349 participants completed the Double-Blind Phase, but did not enter Open-Label Extension Phase.)
Completed | 25 | 20
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- FTC/RPV/TAF: FTC/RPV/TAF (200/25/25 mg) FDC tablet + EFV/FTC/TDF placebo tablet orally once daily for up to 96 weeks.
- EFV/FTC/TDF: EFV/FTC/TDF (600/200/300 mg) FDC tablet + FTC/RPV/TAF placebo tablet orally once daily for up to 96 weeks.
- Total: Total of all reporting groups
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF | Total
Number analyzed (Participants) | 438 | 437 | 875
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48 (9.8) | 47 (10.5) | 48 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 373 | 390 | 763
  Male | 65 | 47 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 9 | 8 | 17
  Black | 118 | 120 | 238
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  White | 291 | 292 | 583
  Not Permitted | 6 | 3 | 9
  Other | 10 | 12 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 78 | 157
  Not Hispanic or Latino | 358 | 359 | 717
  Not Permitted | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 20 | 24 | 44
  Belgium | 3 | 4 | 7
  United States | 351 | 345 | 696
  United Kingdom | 4 | 11 | 15
  France | 7 | 6 | 13
  Switzerland | 6 | 5 | 11
  Germany | 33 | 27 | 60
  Spain | 14 | 15 | 29
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 430 | 432 | 862
  ≥ 50 copies/mL | 8 | 5 | 13
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 711 (292.3) | 688 (263.5) | 700 (278.4)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  ≥ 50 to < 200 cells/µL | 2 | 5 | 7
  ≥ 200 to < 350 cells/µL | 41 | 26 | 67
  ≥ 350 to < 500 cells/µL | 63 | 74 | 137
  ≥ 500 cells/ µL | 332 | 332 | 664

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: The Full Analysis Set included participants who were randomized and received at least 1 dose of study drug and were on EFV/FTC/TDF prior to the screening visit.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 438 | 437
percentage of participants | 90.0 | 92.0
Statistical Analysis 1: Comparison: FTC/RPV/TAF vs EFV/FTC/TDF; The null hypothesis was that the percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 in the FTC/RPV/TAF group was at least 8% lower than the rate in the EFV/FTC/TDF group; the alternative hypothesis was that the percentage of participants with HIV-1 RNA < 50 copies/mL in the FTC/RPV/TAF group was less than 8% lower than that in the EFV/FTC/TDF group; Test type: Non-Inferiority — A sample size of 400 HIV-1 infected participants per treatment group would provide 95% power to detect a non-inferiority margin of 8% in the Week 48 response rate difference between the FTC/RPV/TAF group and EFV/FTC/TDF group. For sample size and power computation, it is assumed that both treatment groups will have a response rate of 89% (based on Gilead Study GS-US-292-0109), that a noninferiority margin is 8%, and that the significance level of the test is at a one-sided alpha level of 0.025; Difference in Percentages = -2.0, 95.001% CI 2-sided [-5.9 to 1.8] — The difference in percentages and its 95.001% confidence interval (CI) were calculated based on an unconditional exact method using 2 inverted 1-sided tests
Statistical Analysis 2: Comparison: FTC/RPV/TAF vs EFV/FTC/TDF; Test type: Superiority; p = 0.35, Fisher Exact

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Defined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 438 | 437
percentage of participants | 1.1 | 0.9

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 96 as Defined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 438 | 437
percentage of participants | 0.7 | 0.9

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96 as Defined by the US FDA-defined Snapshot
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 438 | 437
percentage of participants | 85.2 | 85.1

5. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 390 | 403
cells/µL | 23 (156.4) | 12 (153.3)

6. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 370 | 371
cells/µL | 12 (199.8) | 6 (153.2)

7. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Description: Hip BMD was assessed by dual energy x-ray absorptiometry (DXA) scan.
Time Frame: Baseline; Week 48
Population: Participants in the Hip DXA Analysis Set (all randomized participants received at least 1 dose of study drug, and had nonmissing baseline hip BMD value) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 347 | 367
percentage change | 1.279 (2.3800) | -0.134 (2.4930)

8. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 96
Description: Hip BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Participants in the Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 322 | 345
percentage change | 1.831 (3.2925) | -0.617 (3.3046)

9. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 48
Population: Participants in the Spine DXA Analysis Set (all randomized participants, received at least 1 dose of study drug, and had nonmissing baseline spine BMD values) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 351 | 369
percentage change | 1.645 (3.3198) | -0.045 (2.9087)

10. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 96
Description: Spine BMD was assessed by DXA scan.
Time Frame: Baseline; Week 96
Population: Participants in the Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 327 | 344
percentage change | 1.701 (3.6185) | 0.126 (3.2400)

11. Secondary Outcome: Change From Baseline in HIV Symptoms Index Score (HIVSI) at Week 48
Description: The HIV Symptoms Index was a 20-item, self-reported measure that addressed presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Twenty HIV symptoms including Fatigue, Fever, Dizziness, Hand/Foot Pain, Memory Loss, Nausea, Diarrhea, Sadness, Nervous/anxious, Sleep Trouble, Skin Problems, Cough, Headache, Appetite Loss, Stomach Pain, Muscle/Joint Pain, Sex Problems, Change in Fat Deposits, Weight Loss, and Hair Loss were assessed. There were 5 possible responses (0 = I don't have this symptom; 1 = It doesn't bother me; 2 = It bothers me a little; 3 = It bothers me; and 4 = It bothers me a lot) for each HIV symptom. Total HIV Symptoms Index Score was derived from all 20 HIV symptoms by counting the number of bothersome symptoms. Total score would be missing if any of the individual items were missing.
Time Frame: Baseline; Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 368 | 383
units on a scale | 0 (3.4) | -1 (3.4)

12. Secondary Outcome: Change From Baseline in HIVSI Score at Week 96
Description: as for outcome 11
Time Frame: Baseline; Week 96
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FTC/RPV/TAF | EFV/FTC/TDF
Number analyzed (Participants) | 347 | 347
units on a scale | 0 (4.1) | -1 (3.3)

ADVERSE EVENTS:
Time Frame: First dose date to last dose date (maximum duration: 172.4 weeks) plus 30 days
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- FTC/RPV/TAF (Double-Blind Phase): Adverse events reported occurred during the Double-Blind Phase in participants from the FTC/RPV/TAF group, who received FTC/RPV/TAF (200/25/25 mg) FDC tablet plus EFV/FTC/TDF placebo tablet administered orally once daily.
- EFV/FTC/TDF (Double-Blind Phase): Adverse events reported occurred during the Double-Blind Phase in participants from the EFV/FTC/TDF group, who received EFV/FTC/TDF (600/200/300 mg) FDC tablet plus FTC/RPV/TAF placebo tablet administered orally once daily.
- Open-Label FTC/RPV/TAF From FTC/RPV/TAF: Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Open-Label Extension Phase from the FTC/RPV/TAF group and received FTC/RPV/TAF (200/25/25 mg) FDC tablet once daily.
- Open-Label FTC/RPV/TAF From EFV/FTC/TDF: Adverse events reported occurred during the Open-Label Extension Phase in participants who enrolled into the Open-Label Extension Phase from the EFV/FTC/TDF group and received FTC/RPV/TAF (200/25/25 mg) FDC tablet once daily.
Arm/Group | FTC/RPV/TAF (Double-Blind Phase) | EFV/FTC/TDF (Double-Blind Phase) | Open-Label FTC/RPV/TAF From FTC/RPV/TAF | Open-Label FTC/RPV/TAF From EFV/FTC/TDF
All-Cause Mortality (participants affected / at risk) | 3/438 | 0/437 | 0/25 | 0/21
Serious Adverse Events (participants affected / at risk) | 54/438 | 45/437 | 0/25 | 1/21
Other Adverse Events (participants affected / at risk) | 277/438 | 270/437 | 13/25 | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TAF (Double-Blind Phase) (N=438) | EFV/FTC/TDF (Double-Blind Phase) (N=437) | Open-Label FTC/RPV/TAF From FTC/RPV/TAF (N=25) | Open-Label FTC/RPV/TAF From EFV/FTC/TDF (N=21)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Anal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 0
Bacterial parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis orbital (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis shigella (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Infectious colitis (Infections and infestations) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 3 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 2 | 0 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 3 | 0 | 0
Scrotal infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0
Stoma site abscess (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0
Bipolar II disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 3 | 0 | 0
Fanconi syndrome acquired (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ileostomy closure (Surgical and medical procedures) | 1 | 0 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TAF (Double-Blind Phase) (N=438) | EFV/FTC/TDF (Double-Blind Phase) (N=437) | Open-Label FTC/RPV/TAF From FTC/RPV/TAF (N=25) | Open-Label FTC/RPV/TAF From EFV/FTC/TDF (N=21)
Abdominal pain (Gastrointestinal disorders) | 22 | 13 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 41 | 47 | 1 | 2
Nausea (Gastrointestinal disorders) | 23 | 16 | 0 | 0
Bronchitis (Infections and infestations) | 24 | 28 | 2 | 0
Nasopharyngitis (Infections and infestations) | 51 | 39 | 3 | 1
Pharyngitis (Infections and infestations) | 12 | 19 | 2 | 1
Rhinitis (Infections and infestations) | 5 | 7 | 4 | 0
Sinusitis (Infections and infestations) | 23 | 32 | 1 | 0
Syphilis (Infections and infestations) | 39 | 31 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 74 | 70 | 1 | 1
Urinary tract infection (Infections and infestations) | 22 | 7 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 42 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 37 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 15 | 0 | 0
Headache (Nervous system disorders) | 35 | 31 | 1 | 0
Insomnia (Psychiatric disorders) | 26 | 23 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 30 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 24 | 16 | 0 | 0
Hypertension (Vascular disorders) | 25 | 16 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years